CLINICAL TRIAL: NCT07382895
Title: The Relationship Between the ASA Score Determined by Operating Room Nurses and Intubation Duration
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Zonguldak Ataturk State Hospital (Other)
Responsible Party: Principal Investigator, Tülin KURT ALKAN, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2025-SBB-0079
Record Dates: First submitted 2026-01-12; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: The Individual Must be 18 Years of Age or Older; The Individual Must be Willing to Participate in the Study
Keywords: ASA Physical Status Classification System; preoperative assessment; operating room nurse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Inclusion Criteria for Volunteers in the Study:
  * The person must be 18 years of age or older,
  * The person must be willing to participate in the study.
  Exclusion Criteria for Volunteers in the Study:
  * The person must be 18 years of age or younger,
  * The person must not be a volunteer to participate in the study,
  * The person must be classified as ASA VI,
  * The person must have died during surgery.

SUMMARY:
The objective of this study is to The objective of this study was to ascertain the extent to which operating room nurses assign ASA scores and to assess the reliability of these scores in predicting significant risk factors, including the necessity for mechanical ventilation in patients.

DETAILED DESCRIPTION:
The present research is to be conducted as a prospective observational study. The present prospective observational study is to be conducted over a 3-month period between April 1, 2025, and July 1, 2025, at a single centre, with the involvement of 36 nurses, 12 anesthesiologists (12 operating tables), and 80 patients working in the operating room of Zonguldak Atatürk State Hospital, who evaluate patients in a pre- and post-operative assessment clinic. The sociodemographic information of the nurses and anesthesiologists will be recorded using "Personal Information Form 1" and "Personal Information Form 2". Prior to undergoing surgery, patients' ASA scores and sociodemographic information will be evaluated by operating room nurses and anesthesiologists, who will record this data using "Personal Information Form 3". Patients will be followed up until they are discharged from the clinic, and their mechanical ventilation needs will be recorded. The ASA scores assigned by operating room nurses and anesthesiologists will be analysed in relation to the necessity for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* The person must be 18 years of age or older,
* Must volunteer to participate in the research.

Exclusion Criteria:

* The person must be 18 years of age or younger,
* Not willing to participate in the study,
* The person must be in ASA VI class,
* Death must have been considered during surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was conducted at Zonguldak Atatürk State Hospital between 1 April and 1 July 2025. The operating room was staffed by 36 nurses, 12 anesthesiologists (across 12 operating tables) and 80 patients. A review of extant research on the subject was conducted, and a G Power analysis was subsequently performed. This analysis indicated that, in order to achieve 80% power within a 95% confidence interval for an effect size of d=0.8, it is necessary to include 80 individuals meeting the inclusion criteria in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Determining the sociodemographic information of the nurse using "Personal Information Form 1" | From April 2025 to June 2025
  The nurse's assessment is a nine-item form that includes information such as age, gender, professional work experience, experience working in an operating room, work style, average weekly working hours, income level, and whether or not they have received ASA Physical Status Classification training.
Determining the sociodemographic information of anesthesiologists using "Personal Information Form 3" | From April 2025 to June 2025
  This is an 8-item form that includes the anesthesiologist's age, gender, professional work experience, operating room experience, work style, average weekly working hours, income level, and whether they have received ASA Physical Status Classification training.
Determining the sociodemographic information of the patient's using "Personal Information Form 3" | From April 2025 to June 2025
  This is an 8-item form that includes the patient's age, gender, chronic diseases, previous surgical procedures, Glasgow Coma Scale score, ASA class score, need for mechanical ventilation, and number of days the patient has been intubated.

SECONDARY OUTCOMES:
Comparing patients' ASA scores with their need for mechanical ventilation | From April 2025 to June 2025
  The ASA scores given to patients by operating room nurses and anesthesiologists will be compared with the likelihood of them needing mechanical ventilation. For analyzing the differences between two independent groups with a normal distribution, an independent t-test will be applied; for analyzing the differences between more than two independent groups, an ANOVA test will be applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Atatürk State Hospital, Zonguldak, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patients' personal information was not included in the study and will not be shared.